CLINICAL TRIAL: NCT05711823
Title: ApRepitant in Combination With Granisetron and Dexamethasone versUs Granisetron and dexamEthasone for the Prevention of Vomiting in Patients With HAIC Therapy for Hepatocellular Carcinoma: a Randomized Controlled Study (ARGUE)
Brief Title: Aprepitant Plus Granisetron and Dexamethasone for the Prevention of Vomiting in Patients With HAIC Therapy for HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jian-Hong Zhong, Principal Investigator, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ARGUE
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Aprepitant; Granisetron; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Aprepitant in combination with Granisetron and dexamethasone
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor do not know which patients received antiemetic therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aprepitant in combination with granisetron and dexamethasone (Experimental): Patients with unresectable hepatocellular carcinoma will receive aprepitant in combination with granisetron and dexamethasone during the therapeutic process of hepatic arterial infusion chemotherapy.
  Interventions: Drug: Aprepitant in combination with granisetron and dexamethasone
- granisetron and dexamethasone (Active Comparator): Patients with unresectable hepatocellular carcinoma will receive granisetron and dexamethasone during the therapeutic process of hepatic arterial infusion chemotherapy.
  Interventions: Drug: Granisetron and dexamethasone

INTERVENTIONS:
Drug: Aprepitant in combination with granisetron and dexamethasone — Patients with unresectable hepatocellular carcinoma will receive aprepitant in combination with granisetron and dexamethasone during the therapeutic process of hepatic arterial infusion chemotherapy.
  Arms: Aprepitant in combination with granisetron and dexamethasone
Drug: Granisetron and dexamethasone — Patients with unresectable hepatocellular carcinoma will receive granisetron and dexamethasone during the therapeutic process of hepatic arterial infusion chemotherapy.
  Arms: granisetron and dexamethasone

SUMMARY:
This study aims to evaluate the safety and efficacy of aprepitant combined with granisetron and dexamethasone versus granisetron and dexamethasone in the prevention of nausea and vomiting in patients with hepatocellular carcinoma (HCC) receiving hepatic arterial infusion chemotherapy (HAIC).

DETAILED DESCRIPTION:
FOLFOX regimen include oxaliplatin and 5-Fu. Oxaliplatin has a moderate emetic potential and 5-Fu has a low emetic potential according to European guideline for the prevention of nausea and vomiting caused by chemotherapy and radiotherapy. The Guideline recommend that patients receiving moderately emetogenic chemotherapy receive a three-drug regimen of 5-HT3, dexamethasone, and NK1-RA (aprepitant, fosaprepitant, netupitant or rolapitant). However, HAIC treatment is not through peripheral or central venous infusion of chemotherapy drugs as in other cancers, but through hepatic artery infusion of chemotherapy drugs. Chemotherapy drugs are mainly concentrated in the liver and belong to local chemotherapy, rather than systemic chemotherapy through the venous system. Therefore, although the HAIC regimen includes oxaliplatin and 5-Fu, two chemotherapeutic drugs that may cause vomiting, the literature on whether three-drug regimen is also needed to prevent vomiting has been less publicly reported. In order to further determine whether three-drug regimen is necessary, this project intends to conduct a multi-center, randomized, controlled trial to evaluate the efficacy and safety of aprepitant combined with granisetron and dexamethasone versus granisetron and dexamethasone in preventing nausea and vomiting in HCC patients receiving HAIC treatment. The results of this project will provide a reference for improving the quality of life of HCC patients during HAIC treatment, the compliance of follow-up treatment and saving medical resources.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old;
* The patient is diagnosed with hepatocellular carcinoma according to the clinical diagnostic criteria of the Guideline for Diagnosis and Treatment of Primary Liver Cancer (2022 Edition) issued by the Health Commission of the People's Republic of China or confirmed by histopathology;
* ECOG performance score 0 or 1;
* Child-Pugh score of 5-7 (liver function);
* Receiving hepatic arterial infusion chemotherapy treatment;
* Expected survival time ≥6 months;
* Hematological indexes should meet the following conditions: hemoglobin ≥90 g/L; Absolute neutrophil count ≥1.5×10^9/L; Platelet ≥75×10^9/L; Total bilirubin ≤1.5×ULN; ALT≤3×ULN; AST≤3 x ULN; Alkaline phosphatase (AKP) ≤2.5×ULN; Serum albumin ≥28 g/L; Serum creatinine ≤1.5×ULN;
* Urine protein <2+ or 24h urine protein quantity < 1.0g;
* For women of childbearing age, contraceptive measures (such as intrauterine devices, contraceptive tablets or condoms) are required during the clinical trial until 120 days after the end of the clinical trial; Women of childbearing age had negative serum or urine HCG test results within 7 days prior to study inclusion; Male patients with fertile partners should use effective contraception during the study period and for 120 days after the study ends.

Exclusion Criteria:

* Received systematic chemotherapy in the past;
* The presence of congenital or acquired immunodeficiency diseases (such as HIV positive);
* Active infection, or body temperature ≥ 38.5℃ or white blood cell count > 15 x 10^9/L 7 days before enrollment;
* Complications of arterial or venous thrombosis, such as cerebrovascular accident, deep vein thrombosis and pulmonary infarction, etc. within 6 months;
* Those who have a history of alcohol or psychotropic drug abuse and cannot quit or have mental disorders;
* Pregnant or lactating women;
* being treated with immunosuppressants or glucocorticoids (>10mg prednisone equal dose per day) within 2 weeks;
* Previous history of motion sickness, or combined with hepatic encephalopathy or brain metastases;
* Uncontrolled heart disease or symptoms (including but not limited to grade II or above heart function, unstable angina, myocardial infarction in the past 1 year, supraventricular or ventricular arrhythmias requiring treatment or intervention)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | 3 weeks
  Complete response rate during the first cycle defined as no emetic episodes, no rescue medication use during the first cycle of HAIC therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Le-Qun Li, Study Chair — Guangxi Medical University Cancer Hospital

IPD SHARING:
Plan to Share IPD: No
Data available on request due to privacy/ethical restrictions.

REFERENCES:
- [Background] Zhao Y, He M, Liang R, Li Q, Shi M. Evaluation of Antiemetic Therapy for Hepatic Arterial Infusion Chemotherapy with Oxaliplatin, Fluorouracil, and Leucovorin. Ther Clin Risk Manag. 2021 Jan 22;17:73-77. doi: 10.2147/TCRM.S283192. eCollection 2021. PMID 33519205
- [Background] Roila F, Molassiotis A, Herrstedt J, Aapro M, Gralla RJ, Bruera E, Clark-Snow RA, Dupuis LL, Einhorn LH, Feyer P, Hesketh PJ, Jordan K, Olver I, Rapoport BL, Roscoe J, Ruhlmann CH, Walsh D, Warr D, van der Wetering M; participants of the MASCC/ESMO Consensus Conference Copenhagen 2015. 2016 MASCC and ESMO guideline update for the prevention of chemotherapy- and radiotherapy-induced nausea and vomiting and of nausea and vomiting in advanced cancer patients. Ann Oncol. 2016 Sep;27(suppl 5):v119-v133. doi: 10.1093/annonc/mdw270. No abstract available. PMID 27664248